CLINICAL TRIAL: NCT07351487
Title: Neoadjuvant Chemotherapy Combined With Sintilimab and Bevacizumab for Triple Negative Breast Cancer:A Prospective, Single-Arm, Multicenter Clinical Study (NEOTORCII-BREASTO7)
Brief Title: Neoadjuvant Chemotherapy Combined With Sintilimab and Bevacizumab for TNBC (NEOTORCH-BREAST07)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT20250144C-R1
Record Dates: First submitted 2026-01-12; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-09

CONDITIONS: TNBC - Triple-Negative Breast Cancer
Keywords: TNBC; Sintilimab; Bevacizumab
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — sintilimab; Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant chemotherapy combined with Sintilimab and Bevacizumab (Experimental): 1, Neoadjuvant Chemotherapy Phase Combined with Sintilimab and Bevacizuma, Administered intravenously: carboplatin (AUC=5), nab-paclitaxel (260 mg/m²) + 200 mg Sintilimab + Bevacizumab (7.5 mg/kg), every 3 weeks for a total of 12 weeks. 2, Receive Breast Cancer Definitive Surgery After 4 Cycles of Neoadjuvant Chemotherapy 3, Postoperative Adjuvant Therapy 1)If pathology indicates pCR: Continue immunotherapy, administering 200 mg Sintilimab intravenously every 3 weeks for a total of 1 year. 2)If pathology indicates non-PCR: Continue 4 cycles of postoperative adjuvant chemotherapy (100 mg/m² Epirubicin + 600 mg/m² Cyclophosphamide) combined with 200 mg Sintilimab intravenously every 3 weeks for a total of 1 year. 4, Perform Gene Testing on Biopsy Tissue Before Treatment, and Collect Blood Samples for ctDNA Testing Before and After Treatment.
  Interventions: Drug: Neoadjuvant chemotherapy combined with Sintilimab and Bevacizumab

INTERVENTIONS:
Drug: Neoadjuvant chemotherapy combined with Sintilimab and Bevacizumab — 1, Neoadjuvant Chemotherapy Phase Combined with Sintilimab and Bevacizuma, Administered intravenously: carboplatin (AUC=5), nab-paclitaxel (260 mg/m²) + 200 mg Sintilimab + Bevacizumab (7.5 mg/kg), every 3 weeks for a total of 12 weeks. 2, Receive Breast Cancer Definitive Surgery After 4 Cycles of Neoadjuvant Chemotherapy 3, Postoperative Adjuvant Therapy 1)If pathology indicates pCR: Continue immunotherapy, administering 200 mg Sintilimab intravenously every 3 weeks for a total of 1 year. 2)If pathology indicates non-PCR: Continue 4 cycles of postoperative adjuvant chemotherapy (100 mg/m² Epirubicin + 600 mg/m² Cyclophosphamide) combined with 200 mg Sintilimab intravenously every 3 weeks for a total of 1 year. 4, Perform Gene Testing on Biopsy Tissue Before Treatment, and Collect Blood Samples for ctDNA Testing Before and After Treatment.

SUMMARY:
This study is a prospective, single arm, multi-center phase II clinical trial. The primary study objective is to evaluate the pathologic complete response（PCR） of treatment of TNBC breast cancer with neoadjuvant chemotherapy combined with Sintilimab and Bevacizumab , including the incidences and types of adverse events. The secondary study objective is to observe and evaluate the event-free survival (EFS), Objective Response Rate(ORR), and radiologic complete response (rCR).

ELIGIBILITY:
Inclusion Criteria:

1. Female patients aged 18-70 years old;
2. ECOG score is 0-1 points;
3. Histologically confirmed stage II-III (T1N1-3; T2-4N0-2) invasive breast cancer;
4. ER-negative, PR-negative, and HER2 receptor-negative. Alternatively, if ER and PR expression is less than 10% and HER2 receptor is negative, it is also classified as TNBC;
5. Pathological examination of PD-L1 expression: The Combined Positive Score (CPS) refers to the percentage of PD-L1 positive cells (including tumor cells, lymphocytes, macrophages) in all tumor cells. Our center detected the PD-L1 antibody site as 22C3.
6. The functional level of major organs must meet requirements
7. For female patients who have not yet reached menopause or undergone surgical sterilization: during the treatment period and in the study treatment, the final use effective contraceptive methods for at least 6 months after a single administration.
8. Voluntarily join this study, sign an informed consent form, have good compliance, and are willing to cooperate with follow-up.

Exclusion Criteria:

1. Stage IV breast cancer.
2. Inflammatory breast cancer.
3. Previously received anti-tumor treatment or radiation therapy for any malignant tumor, excluding those that have been cured Malignant tumors such as cervical carcinoma in situ, basal cell carcinoma, or squamous cell carcinoma.
4. Simultaneously undergoing anti-tumor treatment in other clinical trials, including but not limited to chemotherapy and endocrine therapy. Treatment, biological therapy, bone improvement drug therapy, or immune checkpoint inhibitor therapy, etc.
5. The patient had undergone major surgical procedures unrelated to breast cancer within 4 weeks before the first administration of the study drug, or the patient has not fully recovered from such surgical procedures.
6. Serious heart disease or discomfort, including but not limited to the following diseases:

1) Diagnosed history of heart failure or systolic dysfunction (LVEF less than 50%).2) High risk uncontrolled arrhythmias, such as atrial tachycardia, resting heart rate greater than 100bpm, significant ventricular arrhythmias (such as ventricular tachycardia), or higher-level atrioventricular block (i.e. Mobitz II second or third degree atrioventricular block).3) Angina requiring medication for treatment. 4) Heart valve disease with clinical significance. 5) ECG shows transmural myocardial infarction. 6) Poor control of hypertension (systolic blood pressure greater than 180mmHg and/or diastolic blood pressure greater than 180mmHg after drug treatment) 100mmHg).

7. Uncontrolled active infections that require treatment; History of immunodeficiency, including HIV testing positive Sexual, or suffering from other acquired or congenital immunodeficiency diseases, or having a history of organ transplantation.

8. Patients with chronic active hepatitis B or active hepatitis C (excluding hepatitis B virus carriers, stable hepatitis B after drug treatment [HBV-DNA test negative or<50IU/ml] and cured hepatitis C patients [HCV RNA test negative]).

9. Have received immunotherapy and experienced adverse immune events such as immune related pneumonia and myocarditis, which have been determined by researchers to potentially affect the safety of the experimental medication.

10. Individuals with a known history of allergies to the components of this medication regimen.

11. Pregnant and lactating female patients, female patients with fertility and positive baseline pregnancy test results, or reproductive age patients who are unwilling to take effective contraceptive measures during the entire trial period and within 6 months after the last study medication.

12. Suffering from serious accompanying diseases or other comorbidities that may interfere with the planned treatment, or any other circumstances that the researcher deems unsuitable for the patient to participate in this study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2025-09-25 (Actual); Primary Completion 2028-09-25 (Estimated); Study Completion 2030-09-25 (Estimated)

PRIMARY OUTCOMES:
pathologic complete response（PCR） | 3 years

SECONDARY OUTCOMES:
Event free survival (EFS) | 5 years
objective response rate (ORR) | 3 years
radiologic complete response (rCR) | 3 years

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - The First Affiliated Hospital of Anhui Medical University, Hefei
  - Zhongshan Hospital, Fudan University, Shanghai

IPD SHARING:
Plan to Share IPD: No